CLINICAL TRIAL: NCT03393000
Title: Open-label, Randomized, Controlled, Phase 3 Safety and Efficacy Study of Trans Sodium Crocetinate With Radiation Therapy and Temozolomide in Newly Diagnosed Glioblastoma (GBM) Biopsy-Only Subjects
Brief Title: Safety and Efficacy Study of Trans Sodium Crocetinate (TSC) in Newly Diagnosed Glioblastoma (GBM) Biopsy-Only Subjects
Acronym: INTACT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision on behalf of the Sponsor.
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-206
Record Dates: First submitted 2017-12-26; First posted 2018-01-08 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — trans-sodium crocetinate; Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trans Sodium Crocetinate plus SOC (Experimental): Trans Sodium Crocetinate plus the Standard of Care (SOC): SOC composed of radiation and temozolomide for 6 weeks followed by 4 weeks of rest followed by six (6) 28-day cycles of temozolomide
  Interventions: Drug: Trans Sodium Crocetinate plus SOC
- Standard of Care (SOC) (Active Comparator): Standard of Care (SOC): SOC composed of radiation and temozolomide for 6 weeks followed by 4 weeks of rest followed by six (6) 28-day cycles of temozolomide
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Trans Sodium Crocetinate plus SOC — Trans Sodium Crocetinate (TSC) plus the Standard of Care (SOC): SOC composed of radiation and temozolomide for 6 weeks followed by 4 weeks of rest followed by six (6) 28-day cycles of temozolomide
  Other Names: Trans Sodium Crocetinate (TSC) plus Standard of Care
  Arms: Trans Sodium Crocetinate plus SOC
Other: Standard of Care (SOC) — Standard of Care (SOC): SOC composed of radiation and temozolomide for 6 weeks followed by 4 weeks of rest followed by six (6) 28-day cycles of temozolomide
  Other Names: Standard of Care
  Arms: Standard of Care (SOC)

SUMMARY:
Open-label, randomized, controlled, phase 3 safety and efficacy registration trial.

Subjects will be randomized at baseline to the standard of care for first-line treatment of glioblastoma plus Trans Sodium Crocetinate (TSC) or the standard of care.

The standard of care for GBM will consist of temozolomide plus radiation therapy for 6 weeks followed by 28 days of rest followed by 6 cycles of post-radiation temozolomide treatment.

DETAILED DESCRIPTION:
During the radiation treatment period subjects will receive:

1. Focal radiation delivered as 60 Gray/30 fractions scheduled at 2 Gray/day for 5 days each week (Monday through Friday) for 6 weeks.
2. Temozolomide 75mg/m2 orally once daily (usually administered the night preceding each radiation session) starting the evening before the first radiation session over a period of 42 calendar days with a maximum of 49 days.
3. TSC 0.25 mg/kg IV for 3 days each week (Monday, Wednesday, Friday) administered between 45 to 60 minutes prior to each radiation session.

Pneumocystis carinii pneumonia (PCP) prophylaxis is required during Temozolomide + radiation administration, regardless of lymphocyte count and is to continue until recovery of lymphocyte count to less than or equal to Grade 1.

During the 28-day rest period all subjects will receive no treatment.

During the post-radiation 6-cycle temozolomide treatment period subjects will receive:

All subjects will receive: 28-day oral temozolomide (150 mg/m2 first cycle and 200 mg/m2 all subsequent cycles as tolerated) administered on Day 1-5 (Monday through Friday) of each 28-day cycle.

Controls: Will receive oral temozolomide at night at home per the standard of care.

Subjects randomized to TSC: Will receive TSC 1.5 mg/kg (or the dose recommended by the Data Safety Monitoring Board) 1.5 to 2 hours before their temozolomide dose during the daytime for 3 days during the first week of each 28-day cycle (Days 1, 3, 5: Monday, Wednesday, Friday). The Tuesday, Thursday doses will be given at night at home. Long-acting antiemetics may be administered prior to daytime temozolomide dosing on Days 1, 3, 5.

In accordance with the FDA directive of August 22, 2017 the safety, tolerability and pharmacokinetics of TSC at doses between 0.25 mg/kg and up to 1.5 mg/kg in combination with concomitant temozolomide will be assessed via a dose escalation run-in prior to initiating the randomized trial.

The first eight (8) subjects enrolled in the 100-206 trial will be assigned (not randomized between treatments) at Baseline to undergo radiation plus temozolomide plus TSC treatment (0.25 mg/kg) for 6 weekly cycles followed by 4 weeks of rest in standard fashion. At the Week 10 clinic visit the same eight (8) subjects will be assigned to treatment with 2 subjects each assigned to TSC at doses of 0.25, 0.50, 1.0 and 1.5 mg/kg.

The first eight (8) subjects will be studied in parallel and all for two full 28-day cycles with inclusion of appropriate blood sampling collection for TSC and temozolomide pharmacokinetics.

The Data Safety Monitoring Board will examine the resultant safety data after 2 full cycles (Weeks 11 through 18 of post-radiation temozolomide treatment period; Days 1 to 56).

The eight (8) subjects that are a part of the dose-escalation run-in will continue at their assigned TSC dose (0.25, 0.5, 1.0, 1.5 mg/kg) for the Week 19 TSC dosing period.

The Data Safety Monitoring Board will recommend an acceptable TSC dose, if different than 1.5 mg/kg, for the post-radiation temozolomide treatment period prior to the Week 23 TSC dosing period for the eight (8) subjects that are a part of the dose-escalation run-in.

Thereafter, subjects will enter the 100-206 trial and be randomized at Baseline between TSC plus standard of care or the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are at least 18 to 70 years of age
2. Have histologically confirmed GBM
3. The only surgical consideration is biopsy. Subjects who had gross total resection, partial resection and/or debulking are excluded.
4. Measurable (>10mm x 10mm) contrast enhancing disease.
5. Limited disturbance of tumor during biopsy.
6. Surgical and pathology reports that document surgery was limited to biopsy and histologic confirmation.
7. Life expectancy of at least 3 months.
8. Subjects must have a Karnofsky score (KPS) of ≥ 60 at Screening.
9. Glucocorticoid therapy allowed.
10. Tumor Treatment Field (TT Fields) therapy allowed.
11. If female, the subject must have a negative serum or urine pregnancy test at Screening unless meeting non-productive potential criteria.
12. Subjects must have hematologic and renal functions as specified: Absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, Hgb ≥ 9.0g/dL, creatinine ≤ 1.7mg/dL, total bilirubin ≤ 1.5mg/dL, blood urea nitrogen (BUN) within 2 times the upper limit of normal, transaminases ≤ 4 times above the upper limits of the institutional norm.
13. The subject or subject's medical power of attorney has provided written consent to participate in this study.

Exclusion Criteria:

1. Subjects who had gross total tumor resection, partial resection, and/or debulking surgery.
2. Subjects must not have had prior RT, chemotherapy (including Gliadel wafer), immunotherapy or therapy with a biologic agent, or hormonal therapy.
3. Subject who is pregnant or lactating.
4. Subject with a serious concurrent infection or medical illness that would jeopardize the ability of the subject to receive study treatment with reasonable safety.
5. Subject who cannot undergo MRI.
6. Subject receiving concurrent chemotherapeutics or investigational agents within 30 days of study entry, including gliadel wafers or gliasite application.
7. Subjects with other uncontrolled medical conditions, e.g. myocardial infarction, cerebrovascular accident, diabetes or hypertension.
8. Subjects diagnosed with another malignancy within 3 years prior to study start with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma, non-melanomatous skin cancer or carcinoma in situ of the uterine cervix.
9. CTCAE Version 4, Grade 4 non-hematological toxicity (except for alopecia, nausea, vomiting).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry N Cook, RPH/MBA, Study Director — Diffusion Pharmaceuticals Inc
Locations (13):
- United States (13):
  - University of California, Irvine, California
  - Scott Peak, M.D., Redwood City, California
  - John Wayne Cancer Institute @ Providence Saint John's Health Center, Santa Monica, California
  - Piedmont Cancer, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - John Theurer Cancer Center, Hackensack, New Jersey
  - UNM Comprehensive Cancer Center, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Scott Lindhorst, M.D., Charleston, South Carolina
  - Neuro Oncology Associates, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based on the request from FDA for a run-in period prior to initiating the randomized portion of the trial, only the run-in was completed; the randomized trial was never initiated. All results reported are specific to the run-in period.
Period: Overall Study
Arm/Group | Trans Sodium Crocetinate Plus SOC
Started | 19 (23 subjects screened)
Completed | 5 (19 subjects treated)
Not Completed | 14
Not completed — Death | 11
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trans Sodium Crocetinate Plus SOC
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival will be calculated from randomization to the time of death from any cause
Time Frame: All subjects will be followed for 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trans Sodium Crocetinate Plus SOC
Number analyzed (Participants) | 19
Months | 11.3 [5.1 to 19.4]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAE) were recorded if they started or worsened after the first dose of study treatment and within 30 days of the last dose.
Arm/Group | Trans Sodium Crocetinate Plus SOC
All-Cause Mortality (participants affected / at risk) | 14/19
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trans Sodium Crocetinate Plus SOC (N=19)
Cognitive disorder (Nervous system disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Steroid withdrawal syndrome (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Respiratory Syncytial virus infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1)
Intellectual disability (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Vasogenic cerebral oedema (Nervous system disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trans Sodium Crocetinate Plus SOC (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 10
Gait disturbance (General disorders) | 4
Oedema peripheral (General disorders) | 6
Fall (Injury, poisoning and procedural complications) | 4
Aphasia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 7
Vasogenic cerebral oedema (Nervous system disorders) | 4
Confusional state (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6
Deep vein thrombosis (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
The 100-206 trial was an open-label, dose-escalation safety run-in for what was originally planned as a larger randomized trial. 19 pts were enrolled to ensure that at least 8 pts completed the FDA-specified 24-mo. exposure period. At its Q3 2019 meeting, the DSMB found no adverse safety signal and recommended the trial continue as planned. However, the Sponsor did not have resources to fully support the randomized phase of the study and enrollment in the randomized phase was suspended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03393000/Prot_SAP_000.pdf